CLINICAL TRIAL: NCT03568357
Title: Reoxygenation Cardiopulmonary Bypass for Surgical Repair of Pediatric Cyanotic CHD
Brief Title: Reoxygenation for Cyanotic Pediatric CHD
Acronym: Reoxygenation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Clinical Investigator, Peking Union Medical College
Other Study IDs: TedaICH-ROC
Record Dates: First submitted 2017-12-24; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Tetralogy of Fallot
Keywords: tetralogy of Fallot
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Reoxygenation: After one minute of full bypass, fraction of inspired oxygen (FiO2) in liberal group was increased at increments of 0.1 per minute to reach a FiO2 target of 40%-80% adjusted reoxygenation to maintain PO2 in the range of 250mm Hg-300 mm Hg or more during the bypass.
  Interventions: Procedure: Reoxygenation

INTERVENTIONS:
Procedure: Reoxygenation — After one minute of full bypass, fraction of inspired oxygen (FiO2) in conservative group was increased at increments of 0.1 per minute to reach an FiO2 target of 40% that was adjusted to maintain an arterial PO2 in the range of 250 mm Hg or less during the bypass, while FiO2 in liberal group was increased at increments of 0.1 per minute to reach a FiO2 target of 80% adjusted to maintain PO2 in the range of 300 mm Hg or more, on the basis of arterial PO2 level measured via a point of care blood gas analyzer.

SUMMARY:
Evidence is emerging that those patients with cyanotic pathologies may be more vulnerable to end-organ injury during and after surgery than those patients without, because of compromised cardiopulmonary performances or the proinflammatory state that follows conventional hyperoxic cardiopulmonary bypass.

Several clinical and basic studies have identified that controlled oxygenation during the initiation of bypass significantly improved the cardiac adaptation and remodeling capacity than hyperoxic oxygenation strategy among cyanotic patients undergoing tetralogy of Fallot repair, as evidenced by these reduced myocardial gene expression profiles associated with reoxygenation injury.

The investigators designed the reoxygenation for pediatric cardiac surgery study to investigate the effect of reoxygenation during cardiopulmonary bypass on clinical outcomes in patients with cyanotic congenital heart disease .

ELIGIBILITY:
Inclusion Criteria:

* The operation-naive infants and young children aged 1 months to 18 years old were eligible for enrolment if they were indicated for undergoing anticipated radical repair of cyanotic congenital heart disease with cardiopulmonary bypass.

Exclusion Criteria:

* The chromosomal defects, airway and parenchymal lung disease, immunodeficiency, blood transfusion during the current admission, previous cardiac operation, or the opinion of the treating physician that randomization would not be in the best interest of the patient (lack of equipoise)

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The infants and young children aged 1 months to 18 years were eligible for enrolment in this study if they had echocardiography confirmed congenital heart diseases.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Pediatric Logistic Organ Dysfunction (PELOD-2) score | up to 30 days
  the change in the updated Pediatric Logistic Organ Dysfunction (PELOD-2) score (PELOD-2 score; range, 0 to 33 points, with higher scores indicating more severe organ dysfunction)

SECONDARY OUTCOMES:
low cardiac output syndrome | up to 30 days
  Low cardiac output syndrome was defined as cardiac index < 2.2 L/min/m2 of BSA with central venous pressure >18 mmHg and mean arterial pressure < 50 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaocheng Liu, MD, Principal Investigator — TEDA International Cardiovascular Hospital
Locations (1):
- TEDA International Cardiovascular Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babu B, Bhat S, Prabuswamy HP, Kamalapurkar G, Kumar HV, Libu GK, Shilpa S, Lokesh BK. Controlling oxygenation during initiation of cardiopulmonary bypass: can it improve immediate postoperative outcomes in cyanotic children undergoing cardiac surgery? A prospective randomized study. World J Pediatr Congenit Heart Surg. 2012 Jul 1;3(3):310-6. doi: 10.1177/2150135111431843. PMID 23804862
- [Background] Matheis G, Abdel-Rahman U, Braun S, Wimmer-Greinecker G, Esmaili A, Seitz U, Bastanier CK, Moritz A, Hofstetter R. Uncontrolled reoxygenation by initiating cardiopulmonary bypass is associated with higher protein S100 in cyanotic versus acyanotic patients. Thorac Cardiovasc Surg. 2000 Oct;48(5):263-8. doi: 10.1055/s-2000-7879. PMID 11100757
- [Derived] Yang JN, Zhang XM, Ma LY, Lu ZJ, Zheng SQ, Hamzah AW, Shao YF, Liu H, Liu GL. Effect of cardiopulmonary bypass reoxygenation on myocardial dysfunction following pediatric tetralogy of Fallot repair. BMC Cardiovasc Disord. 2021 Apr 26;21(1):210. doi: 10.1186/s12872-021-02033-2. PMID 33902450